CLINICAL TRIAL: NCT03483974
Title: Utilize Hyperspectral Imaging to Reveal the Possible Clues of Neoplasm for Early Stage Detection
Brief Title: Hyperspectral Imaging for Neoplasm Early Stage Detection
Acronym: HINED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Dong-Ru Ho, Assistant Professor, Chang Gung Memorial Hospital
Other Study IDs: 201701068B0
Record Dates: First submitted 2018-03-24; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Hyperspectral Imaging Data of Excreta
Keywords: Hyperspectrum, excreta, neoplasm,
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neoplasm: neoplasm found in follow up
  Interventions: Diagnostic Test: hyperspectral imaging
- non-neoplasm: non-neoplasm patients in follow up
  Interventions: Diagnostic Test: hyperspectral imaging

INTERVENTIONS:
Diagnostic Test: hyperspectral imaging — using hyperspectral detector for evaluation excreta pattern

SUMMARY:
Background Information With the advance in cancer biology, we realize that malignant neoplasm is related with different biological patterns in metabolome and microbiota. Because of the progress in optical spectrometry, it has become possible to evaluate whole visible and innon-visiable absorptive spectrum in human specimens, which may enable detection of minor changes in compound related with altered metabolome and microbiota. We hope to utilize hyperspectral imagingthis spectrum technology to reveal the possible clues of neoplasm for early stage detection

Material and Methods This research intended to enroll one hundred patients into the study. This includes patients with positive stool or urine analysis admitted for workup of colorectal cancer. We will scan the stool and urine with hyperspectral imaging sensoroptical spectrometer, which utilize multichannel charge-coupled device and InGaAs array to analyze the full spectrum of light patterns. The image pattern will be stored and used to linked final diagnosis. Absorption, scattering, and reflection spectra are expected for analysis. Follow up analysis after cancer staging will be used for lowering background noise in all spectra.

Expected Results We expect that there will be specific spectral pattern in stool of colorectal cancer patients, which may be related with cancer staging and different from those in patients without malignancy. Difference in spectra will lead to discovery of new biomarker for colorectal cancer and related diseases. The optic spectra pattern of stool and urine may assist early diagnosis and staging of different malignancies

DETAILED DESCRIPTION:
Background Information With the advance in cancer biology, we realize that malignant neoplasm is related with different biological patterns in metabolome and microbiota. Because of the progress in optical spectrometry, it has become possible to evaluate whole visible and innon-visiable absorptive spectrum in human specimens, which may enable detection of minor changes in compound related with altered metabolome and microbiota. We hope to utilize hyperspectral imagingthis spectrum technology to reveal the possible clues of neoplasm for early stage detection

Material and Methods This research intended to enroll one hundred patients into the study. This includes patients with positive stool or urine analysis admitted for workup of colorectal cancer. We will scan the stool and urine with hyperspectral imaging sensoroptical spectrometer, which utilize multichannel charge-coupled device and InGaAs array to analyze the full spectrum of light patterns. The image pattern will be stored and used to linked final diagnosis. Absorption, scattering, and reflection spectra are expected for analysis. Follow up analysis after cancer staging will be used for lowering background noise in all spectra.

Expected Results We expect that there will be specific spectral pattern in stool of colorectal cancer patients, which may be related with cancer staging and different from those in patients without malignancy. Difference in spectra will lead to discovery of new biomarker for colorectal cancer and related diseases. The optic spectra pattern of stool and urine may assist early diagnosis and staging of different malignancies

ELIGIBILITY:
Inclusion Criteria:

* patients with positive stool or urine analysis
* above 20 year-old
* previous stool or urine analysis negative 8 weeks ago

Exclusion Criteria:

* pregnancy
* active gastrointestinal disease one year ago
* active infection
* having surgery within a year
* underlying active gastrointestinal, urinary tract, and coagulation disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with positive stool or urine analysis who are above 20 year-old
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
neoplasm diagnosis | 6 months after examination
  pathology diagnosis in examination

CONTACTS AND LOCATIONS:
Locations (1):
- Dong-Ru Ho, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No